CLINICAL TRIAL: NCT02432690
Title: A Phase II Clinical Study of BBI503 in Asymptomatic Recurrent Ovarian Cancer Patients With CA-125 Elevation
Brief Title: A Study of BBI503 in Asymptomatic Recurrent Ovarian Cancer Patients With CA-125 Elevation
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Sumitomo Pharma America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BBI503-205GYN-M; BBI503-205GOV-M (Other: Sumitomo Pharma Oncology, Inc.)
Record Dates: First submitted 2015-04-29; First posted 2015-05-04 (Estimated); Results first posted 2022-08-29 (Actual); Last update posted 2023-11-15 (Actual); Status verified 2023-11

CONDITIONS: Cancer; Ovarian Cancer
Keywords: Neoplasms
MeSH Terms: conditions — Neoplasms; Ovarian Neoplasms

ARMS (1):
- Arm A (Experimental)
  Interventions: Drug: BBI503

INTERVENTIONS:
Drug: BBI503 — BBI503 will be administered orally, once daily. Dosing will begin at 200 mg once daily, preferably at bedtime and 2 hours after a meal. Dose modification in case of adverse events is allowed according to the schedule below; Full dose: 200 mg daily, Modification Level-1: 100 mg daily, Modification Level-2: 50 mg daily.
  Other Names: Amcasertib; BB503; BBI-503

SUMMARY:
This was an open-label, single-arm, Phase II study in which amcasertib (BBI503) was administered to adult, asymptomatic patients with recurrent ovarian cancer who had elevated CA-125.

ELIGIBILITY:
Key inclusion criteria:

1. Histological or cytological confirmation of epithelial ovarian, primary peritoneal, or fallopian cancer from any previous time point.
2. Recurrent or relapsed after completion of initial therapy of epithelial ovarian, primary peritoneal, or fallopian cancer from any previous time point (includes completion of surgery with or without postoperative chemotherapy, including maintenance chemotherapy)
3. Elevation of CA-125 according to the following definitions:

   * Patients with an elevated CA-125 before chemotherapy and normalization of CA-125 with/after chemotherapy must show evidence of CA-125 greater than or equal to 2 times the upper limit of normal (ULN) on 2 occasions at least 1 week apart
   * Patients with an elevated CA-125 before cancer chemotherapy, which never normalizes, must show evidence of CA-125 greater than or equal to 2 times the nadir value on 2 occasions at least 1 week apart
   * Patients with CA-125 in the normal range before cancer chemotherapy must show evidence of CA-125 greater than or equal to 2 times the ULN on 2 occasions at least 1 week apart

     * For patients who have received subsequent treatment for recurrent cancer, "chemotherapy" in the above criteria refers to the most recent round of chemotherapy.
4. Patients with a history of ovarian cancer who are asymptomatic and who do not have documented previous CA-125 levels may enroll if the CA-125 is greater than three times the ULN on two occasions, at least one week apart
5. Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) of 0

Key exclusion criteria:

1. Symptoms (other than ≤ grade 1 fatigue, anxiety, depression, or other psychological symptoms) that, in the opinion of the treating oncologist, are a direct result of cancer recurrence. (Examples of symptoms that would preclude enrollment include unintentional weight loss, ≥ grade 2 fatigue, and new abdominal pain unrelated to operative procedures for the ovarian malignancy.)
2. Receiving any other investigational agent that would be considered a treatment for the primary neoplasm. Anti-cancer chemotherapy, radiotherapy, immunotherapy, or investigational agents ≤14 days of first dose of study drug
3. Major surgery ≤28 days before start of treatment
4. History of another primary malignancy with an associated disease-free interval of less than 5 years, except for curatively treated basal cell or squamous cell carcinoma of the skin or in situ cancer of the cervix.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2015-06; Primary Completion 2017-01-02 (Actual); Study Completion 2017-01-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 13 participants who met all inclusion criteria and no exclusion criteria were enrolled and received treatment at 1 clinical site in the United States.
Pre-assignment Details: Participants who died, withdrew consent to survival follow up or were lost to follow up were considered to have completed the study.
Groups:
- Arm A: Participants who were enrolled into the study received amcasertib (BBI503), administered orally, once daily. Dosing began at 200 mg once daily, preferably at bedtime and 2 hours after a meal. Dose modification in case of adverse events was allowed according to following schedule: Full dose: 200 mg daily; Modification Level-1: 100 mg daily; Modification Level-2: 50 mg daily.
Period: Overall Study
Arm/Group | Arm A
Started | 13
Completed | 13
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Arm A
Number analyzed (Participants) | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.6 (9.56)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Not Hispanic or Latino | 12
  Hispanic or Latino | 0
  Not Reported | 0
  Unknown | 0
  Missing | 1
Region of Enrollment [Number; unit: participants]
  United States | 13

OUTCOME MEASURES:

1. Primary Outcome: Disease Control Rate (DCR)
Description: Assessed by the Gynecologic Cancer Intergroup (GCIG) guidelines which incorporate both CA-125 response and Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 (the latter applies to patients who have measurable disease). DCR was defined as the proportion of patients who had an overall response of complete response (CR), partial response (PR), or stable disease (SD).
Time Frame: From the date of first treatment, every 8 weeks, until the date of first documented objective disease progression, up to 24 weeks
Population: Due to a lack of efficacy in the solid tumor indications that were evaluated in early-stage trials of this compound, the entirety of the amcasertib development was discontinued by the sponsor. Analysis of the DCR was not performed since data were not collected.
Arm/Group | Arm A
Number analyzed (Participants) | 0

2. Secondary Outcome: Progression Free Survival (PFS)
Description: The effect of amcasertib (BBI503) on PFS in asymptomatic recurrent ovarian cancer patients with CA-125 elevation
Time Frame: The time from the date of first treatment to the date of first documentation of disease progression or death due to any cause, up to 18 months
Population: Due to a lack of efficacy in the solid tumor indications that were evaluated in early-stage trials of this compound, the entirety of the amcasertib development was discontinued by the sponsor. Analysis of the PFS was not performed since data were not collected.
Arm/Group | Arm A
Number analyzed (Participants) | 0

3. Secondary Outcome: Progression Free Survival (PFS)-6
Description: The effect of amcasertib (BBI503) on PFS at 6 months in asymptomatic recurrent ovarian cancer patients with CA-125 elevation
Time Frame: The time from the date of first treatment to the date of first documentation of disease progression or death due to any cause at 6 months
Population: Due to a lack of efficacy in the solid tumor indications that were evaluated in early-stage trials of this compound, the entirety of the amcasertib development was discontinued by the sponsor. Analysis of the PFS-6 was not performed since data were not collected.
Arm/Group | Arm A
Number analyzed (Participants) | 0

4. Secondary Outcome: Objective Response Rate (ORR)
Description: Assessed by the Gynecologic Cancer Intergroup (GCIG) guidelines which incorporate both CA-125 response and Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 (the latter applies to patients who have measurable disease).
Time Frame: From the date of first treatment, every 8 weeks, until the date of first documented objective disease progression, up to 18 months
Population: Due to a lack of efficacy in the solid tumor indications that were evaluated in early-stage trials of this compound, the entirety of the amcasertib development was discontinued by the sponsor. Analysis of the ORR was not performed since data were not collected.
Arm/Group | Arm A
Number analyzed (Participants) | 0

5. Secondary Outcome: Overall Survival (OS) at 6 Months
Description: Defined as the time from enrollment to death due to any cause.
Time Frame: 4 weeks after the patient has been off study treatment, every 3 months thereafter until death, up to 6 months
Population: Due to a lack of efficacy in the solid tumor indications that were evaluated in early-stage trials of this compound, the entirety of the amcasertib development was discontinued by the sponsor. Analysis of the OS at 6 months was not performed since data were not collected.
Arm/Group | Arm A
Number analyzed (Participants) | 0

6. Secondary Outcome: Number of Patients With Adverse Events
Description: Assessment of safety of amcasertib in participants by reporting of adverse events and serious adverse events
Time Frame: The time from the date of first treatment, while the patient is taking amcasertib, and for 30 days after stopping therapy, an average of 4 months.
Measure: Number; unit: participants
Arm/Group | Arm A
Number analyzed (Participants) | 13
participants | 9

ADVERSE EVENTS:
Time Frame: Serious and Other Adverse Events were assessed from the date of first treatment through 30 days of the last administration of study drug, an average of 4 months. All-Cause Mortality was assessed from the date of first treatment until death, up to 18 months.
Arm/Group | Arm A
All-Cause Mortality (participants affected / at risk) | 3/13
Serious Adverse Events (participants affected / at risk) | 1/13
Other Adverse Events (participants affected / at risk) | 9/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A (N=13)
Blood creatinine increased (Investigations) | 1
Acute kidney injury (Renal and urinary disorders) | 1
Urinary tract obstruction (Renal and urinary disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A (N=13)
Diarrhoea (Gastrointestinal disorders) | 8
Abdominal pain (Gastrointestinal disorders) | 5
Nausea (Gastrointestinal disorders) | 4
Vomiting (Gastrointestinal disorders) | 4
Abdominal pain upper (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Hypoaesthesia oral (Gastrointestinal disorders) | 1
Fatigue (General disorders) | 6
Mucosal inflammation (General disorders) | 2
Decreased appetite (Metabolism and nutrition disorders) | 5
Lymphopenia (Blood and lymphatic system disorders) | 3
Blood creatinine increased (Investigations) | 2
Aspartate aminotransferase increased (Investigations) | 1
Bacterial test positive (Investigations) | 1
Haemoglobin decreased (Investigations) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 2
Back pain (Musculoskeletal and connective tissue disorders) | 1
Dizziness (Nervous system disorders) | 1
Migraine (Nervous system disorders) | 1
Anxiety (Psychiatric disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 1
Urinary tract obstruction (Renal and urinary disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less